CLINICAL TRIAL: NCT00449176
Title: A Randomized Double-Blind, Placebo- and Active-Control, Parallel-arm, Phase III Trial With Controlled Adjustment of Dose to Evaluate the Efficacy and Safety of CG5503 Extended-Release (ER) in Subjects With Moderate to Severe Chronic Low Back Pain
Brief Title: A Study to Evaluate the Effectiveness and Safety of Tapentadol (CG5503) Extended Release (ER) in Patients With Moderate to Severe Chronic Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Grünenthal GmbH (Industry)
Responsible Party: Vice President, Compound Developmen Team Leader, Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR013399; R331333PAI3011 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.)
Record Dates: First submitted 2007-03-16; First posted 2007-03-20 (Estimated); Results first posted 2010-06-24 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; Chronic Pain; Pain Assessment; Tapentadol
MeSH Terms: conditions — Low Back Pain; Chronic Pain | interventions — Tapentadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 001 (Experimental): tapentadol (CG5503) ER 50 100 150 200 250 mg twice daily for 15 weeks
  Interventions: Drug: tapentadol (CG5503) ER
- 002 (Active Comparator): oxycodone CR 10 20 30 40 50 mg twice daily for 15 weeks
  Interventions: Drug: oxycodone CR
- 003 (Placebo Comparator): placebo matching placebo twice daily for 15 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: tapentadol (CG5503) ER — 50, 100, 150, 200, 250 mg twice daily for 15 weeks
  Arms: 001
Drug: oxycodone CR — 10, 20, 30, 40, 50 mg twice daily for 15 weeks
  Arms: 002
Drug: placebo — matching placebo twice daily for 15 weeks
  Arms: 003

SUMMARY:
The purpose of this trial is to evaluate the effectiveness (level of pain control) and safety of orally administrated tapentadol (CG5503) Extended Release (ER) (base) at doses of 100-250 mg twice daily in patients with moderate to severe chronic pain of the lower back, in comparison with placebo and Oxycodone Controlled Release (CR).

DETAILED DESCRIPTION:
The primary objective of this randomized (study medication assigned to patients by chance), double-blind (neither patient nor investigator knows the study medication), phase III, placebo and active controlled trial is to evaluate the efficacy and safety of orally administered tapentadol (CG5503) Extended Release (ER) (base) at doses 100-250 mg twice daily in patients with moderate to severe chronic pain of the lower back. The study is being conducted for registration and approval of tapentadol (CG5503) in the US and outside US. The trial will consist of five periods: screening (to assess eligibility), washout (3-7 days with determination of baseline pain intensity), titration (of dose over 3 weeks to the optimal individual level), maintenance (investigational drug intake for 12 weeks with adjustments allowed), and follow-up (2 weeks post treatment discontinuation). The study hypothesis is that the study drug will be more effective than placebo in reducing patients' pain intensity. The Secondary objectives include the collection of pharmacokinetic (related to how the body uses the drug) information for dose verification. The trial objectives will be assessed by comparing the baseline pain level to the level of week 12 of the maintenance phase. This will be done by looking at the patient's pain diary information. Titrate tapentadol (CG5503) ER (extended release) in 50 mg steps to patient's optimal dose ranging between 100mg and 250mg twice a day; Oxycodone CR (controlled release) 20mg to 50mg twice a day; Placebo (no active ingredients). All doses of trial treatment will be taken orally with or without food, for a maximum timeframe of 15 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Men and non-pregnant, non-lactating women having a diagnosis of Lower Back Pain (LBP) of non-malignant origin present for at least 3 months
* Patients taking analgesic medications for at least 3 months prior to screening and/or dissatisfied with their current therapy
* Patients requiring opioid treatment must be taking daily doses of opioid-based analgesic, equivalent to < 160 mg of oral morphine
* Baseline score of =5 on an 11-point numerical rater scale, calculated as the average pain intensity during the last 3 days prior to randomization.

Exclusion Criteria:

* History of alcohol and/or drug abuse in Investigator's judgement
* History of significant liver insufficiency
* chronic hepatitis B or C, or HIV, presence of active hepatitis B or C within the past 3 months
* Life-long history of seizure disorder or epilepsy
* History of malignancy within past 2 years, with exception of basal cell carcinoma that has been successfully treated
* Uncontrolled hypertension
* Patients with severely impaired renal function
* Patients with moderate to severly impaired hepatic function or with laboratory values reflecting inadequate hepatic function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 981 (Actual)
Dates: Start 2007-02; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Etropolski M, Kuperwasser B, Flugel M, Haufel T, Lange B, Rauschkolb C, Laschewski F. Safety and tolerability of tapentadol extended release in moderate to severe chronic osteoarthritis or low back pain management: pooled analysis of randomized controlled trials. Adv Ther. 2014 Jun;31(6):604-20. doi: 10.1007/s12325-014-0128-6. Epub 2014 Jul 2. PMID 24985410
- [Derived] Biondi DM, Xiang J, Etropolski M, Moskovitz B. Evaluation of blood pressure and heart rate in patients with hypertension who received tapentadol extended release for chronic pain: a post hoc, pooled data analysis. Clin Drug Investig. 2014 Aug;34(8):565-76. doi: 10.1007/s40261-014-0209-y. PMID 24916058
- [Derived] Etropolski M, Lange B, Goldberg J, Steup A, Rauschkolb C. A pooled analysis of patient-specific factors and efficacy and tolerability of tapentadol extended release treatment for moderate to severe chronic pain. J Opioid Manag. 2013 Sep-Oct;9(5):343-56. doi: 10.5055/jom.2013.0177. PMID 24353047
- [Derived] Merchant S, Provenzano D, Mody S, Ho KF, Etropolski M. Composite measure to assess efficacy/gastrointestinal tolerability of tapentadol ER versus oxycodone CR for chronic pain: pooled analysis of randomized studies. J Opioid Manag. 2013 Jan-Feb;9(1):51-61. doi: 10.5055/jom.2013.0147. PMID 23709304
- [Derived] Afilalo M, Morlion B. Efficacy of tapentadol ER for managing moderate to severe chronic pain. Pain Physician. 2013 Jan;16(1):27-40. PMID 23340531
- See also: A Study to Evaluate the Effectiveness and Safety of Tapentadol (R331333) Extended Release (ER) in Patients with Moderate to Severe Chronic Low Back Pain — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=68&filename=CR013399_CSR.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period for this out-patient, multicenter study occurred between 21 February 2007 and 12 March 2008.
Pre-assignment Details: The study consisted of a screening period (duration up to 14 days), a washout period (duration 3 to 7 days), a double-blind active treatment period with titration period (duration 3 weeks) and maintenance period (duration 12 weeks).
Groups:
- Tapentadol ER: Tapentadol (CG5503) extended release(ER) 100-250mg twice daily(BID)
- Oxycodone CR: oxycodone controlled release(CR) 20-50mg twice daily(BID)
- Placebo: Matching Placebo twice daily(BID)
Period: Overall Study
Arm/Group | Tapentadol ER | Oxycodone CR | Placebo
Started | 318 (3 randomly assigned to this treatment group did not take drug (of 321 subjects initially randomized)) | 328 (6 randomly assigned to this treatment group did not take drug (of 334 subjects initially randomized)) | 319 (5 randomly assigned to this group did not receive drug, 2 enrolled twice(of 326 subjects randomized))
Completed | 166 | 133 | 152
Not Completed | 152 | 195 | 167
Not completed — Withdrawal by Subject | 39 | 43 | 59
Not completed — Lost to Follow-up | 13 | 8 | 12
Not completed — Adverse Event | 51 | 107 | 15
Not completed — Lack of Efficacy | 13 | 7 | 50
Not completed — Study drug non-compliant | 14 | 11 | 11
Not completed — all other | 22 | 19 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tapentadol ER | Oxycodone CR | Placebo | Total
Number analyzed (Participants) | 318 | 328 | 319 | 965
Age Continuous [Mean (Standard Deviation); unit: years] | 49.4 (13.21) | 50.0 (14.21) | 50.4 (14.05) | 49.9 (13.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 194 | 181 | 184 | 559
  Male | 124 | 147 | 135 | 406

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of the Average Pain Intensity Based on a 11-point Numerical Rating Scale (NRS) Over the Last Week of the Maintenance Period at Week 12.
Description: For this twice daily pain assessment, the subjects were to indicate the level of pain experienced over the previous 12 hours on an 11-point Numerical Rating Scale (NRS) where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine".
Time Frame: Baseline and 12 weeks
Population: Intent To Treat (ITT) analysis set utilizing Last Observation Carried Forward (LOCF) imputation. The ITT analysis set included all randomized patients that took at least one dose of study medication following randomization. 7 patients (3 tapentadol ER, 3 oxycodone CR, 1 placebo) had no baseline pain scores therefore excluded from the analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Tapentadol ER | Oxycodone CR | Placebo
Number analyzed (Participants) | 312 | 323 | 316
scores on a scale | -2.9 (2.66) | -2.9 (2.52) | -2.1 (2.33)
Statistical Analysis 1: Comparison: Tapentadol ER vs Placebo; The primary null hypothesis to be tested for the study was that the tapentadol ER group was not different from the placebo group for the primary endpoint. Assuming the mean treatment group difference of 0.7 with an SD of 2.7, 314 subjects per treatment group were estimated to provide 90% power to show that the tapentadol ER group was statistically different from placebo at an alpha level of 0.05. The total number of subjects to be randomly assigned to a treatment group for the study was 942; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -0.8, 95% CI [-1.22 to -0.47], Standard Error of Mean 0.19

2. Secondary Outcome: Change From Baseline in Brief Pain Inventory (BPI) Total Pain Score Over the Last Week of the Maintenance Period at Week 12.
Description: Total pain score where zero equals "no pain" to ten equals "pain as bad as you can imagine" from 12 week endpoint vs baseline.
Time Frame: Baseline and 12 week endpoint
Population: Intent to Treat (ITT) analysis set, last observation carried forward (LOCF) imputation. The ITT analysis set included all randomized patients that took at least one dose of study medication following randomization. The patients who didi not have any assessment during the treatment period were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Tapentadol ER | Oxycodone CR | Placebo
Number analyzed (Participants) | 314 | 323 | 314
scores on a scale | -2.3 (2.25) [-1.06 to -0.37] | -2.1 (2.35) [-0.88 to -0.2] | -1.6 (2.11)

3. Secondary Outcome: Change From Baseline in Sleep Latency Time in Hours Over the Last Week of the Maintenance Period at Week 12.
Description: A Sleep Questionnaire addressed the following question: "How long after bedtime/lights out did you fall asleep last night (hours)?" 12 week endpoint-mean changes from baseline at endpoint for sleep latency. Decrease in time(hours) indicates improvement.
Time Frame: Baseline and 12 week endpoint
Population: Intent to Treat population with LOCF imputation. The patients who didi not have any assessment during the treatment period were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Tapentadol ER | Oxycodone CR | Placebo
Number analyzed (Participants) | 311 | 324 | 312
hours | -0.2 (3.08) | -0.2 (2.32) | -0.1 (2.43)

4. Secondary Outcome: Percentage of Patients Who Reported Very Much Improved or Much Improved From Baseline in Patient Global Impression of Change Over the Last Week of the Maintenance Period at Week 12
Description: Ordinal measure indicating change from start of treatment (On a scale of 7 = Very much Worse to 1 = very much improved)
Time Frame: Baseline and 12 week endpoint
Population: Intent to Treat Analysis (ITT) set, Last Observation Carried Forward (LOCF) imputation method. The ITT analysis set included all randomized subjects who took at least one dose of study medication following randomization. The patients who didi not have any assessment during the treatment period were excluded from the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Tapentadol ER | Oxycodone CR | Placebo
Number analyzed (Participants) | 236 | 210 | 245
percentage of participants | 55.5 | 60 | 32.7

5. Secondary Outcome: Number of Participants With Treatment Discontinuation Due to Lack of Efficacy
Description: The number of participants who discontinued due to lack of efficacy from baseline to endpoint
Time Frame: Baseline and 12 weeks
Population: Intent to Treat Analysis Set
Measure: Number; unit: participants
Arm/Group | Tapentadol ER | Oxycodone CR | Placebo
Number analyzed (Participants) | 315 | 326 | 317
participants | 18 | 9 | 64 [lower limit 33]

6. Secondary Outcome: Change From Baseline in EuroQol-5® (EQ-5D) Health Status Index to Week 12
Description: Change from baseline to end point in EuroQol-5 Dimension Questionnaire. A higher score indicates an improvement in health in the Health Status Index. The EuroQol-5 is a five dimensional health state classification. Each dimension is assessed on a 3-point ordinal scale (1=no problems, 2=some problems, 3=extreme problems). The responses to the five EQ-5D dimensions were scored using a utility-weighted algorithm to derive an EQ-5D health status index score between 0 to 1, with 1.00 indicating "full health" and 0 representing dead.
Time Frame: Baseline and 12 week endpoint
Population: Intent to Treat Analysis Set, LOCF imputation method. The patients who didi not have any assessment during the treatment period were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Tapentadol ER | Oxycodone CR | Placebo
Number analyzed (Participants) | 315 | 325 | 316
scores on a scale | 0.2 (0.3) | 0.2 (0.33) | 0.1 (0.33)

7. Secondary Outcome: Responder Analysis 50% Improvement
Description: Defined by the proportion of subjects achieving at least 50% improvement from baseline in the primary endpoint of change from baseline of the average pain intensity based on the 11-point Numerical Rating Scale (NRS) at week 12. The subjects were to indicate the level of pain experienced over the previous 12 hours on an 11-point NRS where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine".
Time Frame: Baseline and Week 12
Population: Intent to Treat Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | Tapentadol ER | Oxycodone CR | Placebo
Number analyzed (Participants) | 315 | 326 | 317
Percentage of participants | 27.0 | 23.3 | 18.9

ADVERSE EVENTS:
Time Frame: All adverse events were reported from the time a signed and dated informed consent was obtained throughout the follow-up phase of the study. Serious adverse events were collected for 30 days after the last dose of study drug.
Arm/Group | Tapentadol ER | Oxycodone CR | Placebo
Serious Adverse Events (participants affected / at risk) | 8 | 11 | 3
Other Adverse Events (participants affected / at risk) | 192/318 | 240/328 | 118/319
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Tapentadol ER | Oxycodone CR | Placebo
Abdominal Pain (Gastrointestinal disorders) | 1/318 | 0/328 | 0/319
Anemia (Blood and lymphatic system disorders) | 0/318 | 1/328 | 0/319
Angina Pectoris (Cardiac disorders) | 0/318 | 1/328 | 0/319
Atrial Fibrillation (Cardiac disorders) | 1/318 | 0/328 | 0/319
Bipolar Disorder (Psychiatric disorders) | 0/318 | 0/328 | 1/319
Bladder Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/318 | 1/328 | 0/319
Cardiac Pacemaker Replacement (Surgical and medical procedures) | 1/318 | 0/328 | 0/319
Chest Pain (General disorders) | 0/318 | 1/328 | 0/319
Clostridial Infection (Infections and infestations) | 2/318 | 1/328 | 1/319
Confusional State (Psychiatric disorders) | 1/318 | 0/328 | 0/319
Coronary Artery Bypass (Surgical and medical procedures) | 0/318 | 1/328 | 0/319
Coronary Artery Occlusion (Cardiac disorders) | 0/318 | 1/328 | 0/319
Dehydration (Metabolism and nutrition disorders) | 0/318 | 1/328 | 0/319
Depressed Level of Consciousness (Nervous system disorders) | 1/318 | 0/328 | 0/319
Dizziness (Nervous system disorders) | 0/318 | 1/328 | 0/319
Duodenal Ulcer (Gastrointestinal disorders) | 0/318 | 0/328 | 1/319
Foot Fracture (Injury, poisoning and procedural complications) | 1/318 | 0/328 | 0/319
Gastroenteritis (Infections and infestations) | 1/318 | 1/328 | 0/319
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 0/318 | 1/328 | 0/319
Injury (Injury, poisoning and procedural complications) | 1/318 | 0/328 | 0/319
Non Cardiac Chest Pain (General disorders) | 0/318 | 0/328 | 1/319
Palpitations (Cardiac disorders) | 0/318 | 1/328 | 0/319
Pneumonia (Infections and infestations) | 0/318 | 0/328 | 1/319
Schizoaffective Disorder (Psychiatric disorders) | 0/318 | 1/328 | 0/319
Schizophrenia (Psychiatric disorders) | 0/318 | 0/328 | 1/319
Suicidal Ideation (Psychiatric disorders) | 0/318 | 0/328 | 1/319
Tinnitus (Ear and labyrinth disorders) | 0/318 | 1/328 | 0/319
Transient Ischemic Attack (Nervous system disorders) | 0/318 | 1/328 | 0/319
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tapentadol ER (N=318) | Oxycodone CR (N=328) | Placebo (N=319)
Constipation (Gastrointestinal disorders) | 44 | 88 | 16
Diarrhea (Gastrointestinal disorders) | 19 | 8 | 23
Dizziness (Nervous system disorders) | 38 | 55 | 18
Dry Mouth (Gastrointestinal disorders) | 26 | 12 | 7
Dyspepsia (Gastrointestinal disorders) | 16 | 6 | 8
Fatigue (General disorders) | 21 | 24 | 13
Headache (Nervous system disorders) | 63 | 55 | 44
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 12 | 17 | 0
Insomnia (Psychiatric disorders) | 13 | 25 | 9
Nausea (Gastrointestinal disorders) | 64 | 113 | 29
Pruritus (Skin and subcutaneous tissue disorders) | 23 | 55 | 6
Somnolence (Nervous system disorders) | 42 | 53 | 8
Vomiting (Gastrointestinal disorders) | 29 | 63 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less